CLINICAL TRIAL: NCT01994694
Title: Risk Perception in Adults With Attention Deficit and Hyperactivity Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: riskperception.ctil
Record Dates: First submitted 2013-11-17; First posted 2013-11-26 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-07

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- adults with ADHD: adults with ADHD, without neurological and psychiatric comorbidities
- controls: people without ADHD, with no neurological and psychiatric disorders

SUMMARY:
People with ADHD often engage in risky behaviors, such as dangerous driving, substance abuse and gambling. Current behavioral economy theories differentiate between risk perception and risk attitude. This study aims to measure both risk taking and risk perception in adults with and without ADHD. It is hypothesized that people with ADHD show decreased risk perception, accounting for their risky behavior. In contrast, it is hypothesized that people with ADHD do not show increased risk attitude, namely, they are not risk seeking.

DETAILED DESCRIPTION:
INTRODUCTION:

People with ADHD are found to be engaged in risky behavior and tend to take risks such as dangers driving, substance abuse, gambling and more. These tendencies are in line with findings of poor decision making in individuals with ADHD. Even though none of the existing theories of ADHD manage to explain the full spectrum of decision making among ADHD, yet this population interpreted as risk seekers regardless causative correlation that link the disorder to risk taking behavior. Studies regarding decision making under uncertainty have uncovered common patterns of behavior that are inconsistent with the grasp that individuals with ADHD are risk seekers. First, studies that used gambling tasks showed that subjects with ADHD bet on smaller wages than non ADHD subjects. Second, when subjects with ADHD confronted with risky options that showed similarity in its expected value or that the expected value was beneficial compared to the safe one, they did not choose the risky options. Surprisingly, when the risky options did not carry any gain or benefit they tend to choose the risky options upon the beneficial or safer ones. Third, subjects with ADHD who preformed explicit pure risk seeking tasks under two conditions, with and without feedback, differ from control group only in the with feedback condition and were conservative in choosing risky alternatives. All of the above questions upon the risk perception of people with ADHD in more skeptical light and is being researched in this study in a direct and more comprehensive way.

METHODS:

Participants:

Two hundred adults with and with out ADHD will be recruited through addressing to undergraduate students at the Hebrew University and Talpiot Collage in Israel, who will be enrolled in special education course for teachers, and through addressing work colleagues.

All participants will complete the following questionnaire:

ADHD Adult Self Report Scale (ASRS-v1.1) in order to measure the severity of ADHD symptoms.

Domain-specific Risk-Taking (DOSPERT): The subjects will be asked to complete a paper-and-pencil questionnaire in groups of 5-10 individuals or in private.of the DOSPERT questionnaire consisted of a total set of 30 items assessing 3 scales (risk taking, risk perception and expected benefits) in five domains of risk: financial, health/safety, recreational, ethics, and social, 6 items in each domain. The set of 30 items was presented three times in counterbalanced order.

The Hebrew version of the DOSPERT scale was developed for this study using the method of back-translation. Internal consistency for the 3 measures was good. Cronbach's alpha was 0.85, 0.83 and 0.86, for Risk Taking, Risk Perception and Expected Benefit perception, respectively.

Hypothesis:

We predict that: (a) higher level of ADHD symptoms will be associated with higher risk taking ; (b) lower risk perception and higher benefit perception will be associated with higher risk taking ; (c) higher level of ADHD symptoms will be associated with lower risk perception and higher benefit perception ; (d) risk and benefit perceptions will mediate the relation between level of ADHD symptoms and risk taking.

Analysis:

Three measures will be analyzed: Risk Taking (defined as the willingness to engage in a risky activity as a function of its perceived riskiness), Risk Perception (defined as the reported level of risk taking), and Expected Benefits (define as the benefit responders expect to obtain from engaging in each risky behavior). Correlations with the ASRS scores will be examined. A mediation analysis will be conducted in order to examine the role of risk and benefit perception as potential mediator of ADHD-related risk taking.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of ADHD

Exclusion Criteria:

* any neurological disorder
* any psychiatric disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with ADHD
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Domain-specific Risk-Taking questionnaire | 1 day
  Subjects are given the questionnaire once

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Pollak, PhD, Principal Investigator — Hebrew University of Jerusalem
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel, Israel